CLINICAL TRIAL: NCT05821400
Title: Cognitive Changes in Mild Cognitive Impairment Without Orthostatic Hypotension
Brief Title: Cognitive Changes in Mild Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort-MCI
Record Dates: First submitted 2022-09-29; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Healthy Controls Without Orthostatic Hypotension
Keywords: cognition
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy controls without orthostatic hypotension
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Background: In recent years, the changes of cognitive function in mild cognitive impairment have attracted attention.

Methods/design: We will follow up at 3. The primary outcome will be the measurement of cognitive function using neuropsychological assessment scales such as MOCA, MMSE, etc... Minor variables will be included plasma biomarkers (Aβ, Tau, GFAP, etc.), multimodal brain electrophysiology (P300, VP300, heart rate variability, etc.), and neuroimaging indicators (NODDI).

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed mild cognitive impairment

Exclusion Criteria:

* Patients with orthostatic hypotension
* Patients with other neurological disorders.
* Pregnant or lactating women.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese who met the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Montreal Cognitive Assessment (MoCA) scores after 3 months. | Participants will be followed up for 3 months after baseline.
  The MOCA scale scores range from 0 to 30, with higher scores indicating better cognition

SECONDARY OUTCOMES:
Changes in Plasma amyloid protein levels after 3 months. | Participants will be followed up for 3 months after baseline.
  Plasma amyloid protein(ug/ml) is an important indicator of cognitive function.
Changes in Plasma tau levels after 3 months. | Participants will be followed up for 3 months after baseline.
  Plasma tau(ug/ml) is an important indicator of cognitive function
Changes in Blood pressure (mmHg) after 3 months. | Participants will be followed up for 3 months after baseline.
  An experienced physician will measure blood pressure on the right upper arm after the subject rest for 5 min, taking the average of the two measurements as the final result.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Petersen RC, Roberts RO, Knopman DS, Geda YE, Cha RH, Pankratz VS, Boeve BF, Tangalos EG, Ivnik RJ, Rocca WA. Prevalence of mild cognitive impairment is higher in men. The Mayo Clinic Study of Aging. Neurology. 2010 Sep 7;75(10):889-97. doi: 10.1212/WNL.0b013e3181f11d85. PMID 20820000
- [Background] Rabe-Jablonska J, Bienkiewicz W. [Anxiety disorders in the fourth edition of the classification of mental disorders prepared by the American Psychiatric Association: diagnostic and statistical manual of mental disorders (DMS-IV -- options book]. Psychiatr Pol. 1994 Mar-Apr;28(2):255-68. Polish. PMID 8208869